CLINICAL TRIAL: NCT07329010
Title: The Effect of Preoperative Whey Protein and Physical Exercise Support on Recovery After Total Hip Arthroplasty
Brief Title: Effects of Preoperative Whey Protein and Exercise Support on Recovery After Total Hip Arthroplasty
Acronym: THA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, HÜMEYRA YÜKSEL, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 010203
Record Dates: First submitted 2025-12-02; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Arthoplasty; Nutrition; Geriatric Assessment; Exercise Training; Preoperative
Keywords: Whey Protein; Exercise; Preoperative Nutrition; Total Hip Arthroplasty (THA); Elderly Patients; Postoperative Recovery; Functional Outcomes
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the intervention group, which receives 14 days of preoperative whey protein supplementation combined with a home-based exercise program, or the control group, which receives standard preoperative care. Both groups are followed for metabolic and functional outcomes on postoperative days 3 and 5
Masking Description: This is an open-label study. Neither participants nor investigators are blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: "Preoperative Whey Protein Supplementation and Exercise Program (Experimental): The preoperative exercise and protein supplementation program will be conducted by patients in their home environment. Patients will be enrolled in the study 14 days prior to the scheduled surgery. At the start of the program, all patients will receive face-to-face instructions, and data will be collected under the supervision of an experienced orthopedic surgeon at the hospital
  Interventions: Dietary Supplement: Preoperative Whey Protein and Exercise Program
- Control Group: "Standard Preoperative Care" (No Intervention): Patients in the control group will receive only the hospital's standard preoperative care protocol. This care includes:
  Daily monitoring of vital signs
  Preoperative laboratory tests
  Anesthesia pre-assessment
  Surgical information and counseling
  Medication management
  No additional protein supplementation or exercise training will be provided specifically to this group.

INTERVENTIONS:
Dietary Supplement: Preoperative Whey Protein and Exercise Program — The intervention group will receive 14 days of preoperative whey protein supplementation combined with a home-based exercise program. Patients will receive face-to-face instructions at program initiation, and data will be collected under the supervision of an experienced orthopedic surgeon
  Other Names: Dietary Supplement + Behavioral (Exercise)
  Arms: Intervention Group: "Preoperative Whey Protein Supplementation and Exercise Program

SUMMARY:
Objective:

The aim of this project is to evaluate the effects of preoperative whey protein supplementation and a physical exercise program on postoperative recovery outcomes in patients undergoing total hip arthroplasty (THA). Specifically, inflammatory markers (CRP), nutritional status (albumin), mobilization time, length of hospital stay, and physical and social functioning will be assessed. As one of the first randomized controlled trials in Turkey to focus on the preoperative period and to evaluate a combined nutrition and exercise intervention in elderly surgical patients, this study holds pioneering significance in both clinical and academic contexts.

Methods:

This study is designed as a randomized controlled trial. The intervention group will receive whey protein supplementation and a home-based exercise program for 14 days preoperatively, while the control group will receive standard preoperative care. Data collection will be performed preoperatively and on postoperative days 3 and 5, focusing on metabolic and functional parameters.

Expected Outcomes:

The findings of this study are expected to contribute to the improvement of patient care through a multidisciplinary approach, inform health policy development, and provide a foundation for larger-scale clinical research in Turkey.

DETAILED DESCRIPTION:
Background:

Hip osteoarthritis (HOA) is a common degenerative disease in older adults that leads to pain, deformity, and functional loss, thereby reducing quality of life. Muscle atrophy, neuromuscular dysfunction, and pain are frequently observed in the affected limb, resulting in decreased muscle strength. Gait analyses have shown reduced hip range of motion (ROM), decreased walking speed, and diminished hip flexion and abduction moments.

Total hip arthroplasty (THA), widely used in the treatment of HOA, is also performed for femoral fractures, arthritis, developmental hip dysplasia, and osteonecrosis. Although THA is an effective surgical method, delayed wound healing, infection risk, muscle weakness, and mobilization limitations remain important postoperative challenges. With postoperative pain reduction, hip function and quality of life improve significantly. However, diminished proprioception may cause balance problems, increasing the risk of falls.

Exercise therapy plays a key role in postoperative rehabilitation after THA. Physiotherapists provide gait training, ROM exercises, and balance activities. Exercise therapy reduces pain and increases physical activity levels. Systematic reviews have demonstrated the positive effects of exercise on muscle strength and gait performance following THA.

Nevertheless, delayed wound healing, infection, increased morbidity and mortality, and prolonged hospitalization may still occur after THA. In this context, preoperative nutritional support plays a critical role in improving patient outcomes. Protein-based supplements can support muscle protein synthesis and accelerate recovery. Increased protein intake helps prevent muscle breakdown and supports recovery. Thus, selecting an appropriate nutritional and exercise strategy is essential in the postoperative management of orthopedic patients.

Whey protein (WP) is a protein source rich in branched-chain amino acids (BCAAs) and essential amino acids, with high bioavailability and easy digestibility. WP has been shown to stimulate muscle protein synthesis, enhance recovery, and reduce postoperative infection risk.

In Turkey, the surgical needs of the elderly population are steadily increasing, and THA procedures are becoming a major healthcare requirement, especially in older age groups. While the separate effects of exercise and protein supplementation on postoperative outcomes have been demonstrated, there is no study in Turkey evaluating the combined impact of these two interventions when applied in the preoperative period.

This project aims to be the first randomized controlled trial in elderly THA patients to investigate the effects of oral whey protein supplementation combined with a preoperative exercise program on metabolic markers, early mobilization, and length of hospital stay. Both interventions are safe, cost-effective, and easy to apply, and they allow elderly patients to continue daily activities without additional effort or time burden. This project is expected to contribute significantly to the literature by offering an innovative approach in postoperative THA management and by generating scientific evidence on the interaction between nutrition, exercise, and surgical outcomes. The study will be conducted under the supervision of an experienced orthopedic surgeon, with methodological and practical support from clinical dietitians and physiotherapists. The intervention design, data collection, and analysis procedures are planned in accordance with the literature and scientific standards.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 70 years
* Scheduled for elective total hip arthroplasty (THA)
* Able to participate in the preoperative intervention for at least 2 weeks
* Conscious and able to communicate

Exclusion Criteria:

* Patients with advanced malnutrition
* Patients with active cancer, malabsorption, liver or kidney failure
* Patients with severe cognitive impairment
* Patients with health conditions that prevent participation in exercise

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Serum Albumin Level | 5 days
  Postoperative serum albumin levels measured on days 3 and 5 after total hip arthroplasty.
C-Reactive Protein (CRP) Level | 5 days
  Postoperative serum CRP levels measured on days 3 and 5 after total hip arthroplasty.

SECONDARY OUTCOMES:
Time to Mobilization | 5 days
  Time (in hours) from surgery completion to first independent mobilization.
Length of Hospital Stay | 5 days
  Total duration of hospital stay (in days) after surgery.
Physical and Social Functioning | 5 days
  Assessment of patients' physical and social functioning using standardized scales.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adebero T, Omana H, Somerville L, Lanting B, Hunter SW. Effectiveness of prehabilitation on outcomes following total knee and hip arthroplasty for osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Disabil Rehabil. 2024 Dec;46(24):5771-5790. doi: 10.1080/09638288.2024.2313128. Epub 2024 Feb 13. PMID 38349251